CLINICAL TRIAL: NCT00979810
Title: Image-Guided Stereotactic Biopsy of High Grade Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-060; R21CA137896-01A1 (NIH)
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-02

CONDITIONS: Brain Cancer; Glioma
Keywords: PET scan; CT scan; 09-060; CNS
MeSH Terms: conditions — Brain Neoplasms; Glioma

ARMS (1):
- 18F-FLT PET scan (Experimental): This is a pilot study intended to collect preliminary data on 15 patients diagnosed with untreated high-grade glioma who are scheduled to undergo surgical resection.
  Interventions: Drug: 18F-FLT PET Scan

INTERVENTIONS:
Drug: 18F-FLT PET Scan — The patient will undergo MRI and 18F-FLT PET scans of the brain. A IV catheter will be placed in a superficial hand or arm vein for administration of 18F-FLT (approximately 370 MBq), prepared by the MSKCC Radiochemistry Core Facility. A second venous catheter will be placed in the opposite hand or arm for venous blood sampling. If a central venous catheter is present, it will be used for blood sampling or radiopharmaceutical administration, and only a single venous catheter will be placed. Sequential blood samples may be obtained following 18F-FLT infusion for assaying whole blood and plasma radioactivity. All catheters will be removed at the end of the day.
  Other Names: As part of the standard surgical care for brain cancer, the patient will undergo; biopsy of the tumor. A few small tissue samples will be collected from different; sites within the tumor and used for examining the biology of the tumor tissue.; Associations will be made between the 18F-FLT imaging findings at these biopsy; sites, which reflect differences in tumor growth rate, and the corresponding; biology of the tumor measured in the sampled tumor tissue.

SUMMARY:
The purpose of this study is to evaluate high and low areas of growth, or proliferation, within the tumor. An imaging technique using a very small amount of a radioactive tracer called 18Ffluoro-deoxy-L-thymidine (18F-FLT) can detect areas of rapid growth within the tumor. This imaging technique is called a FLT PET imaging. This present study involves obtaining one scan using FLT PET imaging. The goal of this study is to investigate associations between the imaging findings showing differences in growth rate within the tumor and the biology of the tumor that is measured in the sampled tumor tissue. This information may be used in future brain tumor patients to determine the best combination of treatment for individual patients. These studies may also improve our understanding of the types of changes taking place in brain tumor tissue that could improve individual patient outcome. FLT is produced for human use by the MSKCC cyclotron facility under an investigational new drug (IND) approval issued by the US Food and Drug Administration (FDA). This means that FLT is produced under strict rules and regulations, is considered safe, and has been approved for use in humans for certain disease conditions. 18F-FLT has been used in several research studies to date at this institution.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = to 18 years old.
* Radiographic appearance of a lesion presumed to be high-grade glioma.
* Planned surgical resection.

Exclusion Criteria:

* All patients who have been previously treated with radiation, chemotherapy, or other targeted drugs (patients only) for their brain tumor.
* Pregnant (confirmed by serum b-HCG in women of reproductive age) or breast feeding.
* Patients with other active malignancies or prior treatment for non-CNS malignancies.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09-16 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Bradbury, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 18F-FLT PET Scan
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18F-FLT PET Scan
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 57 [41 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Invest Relation Btw Voxel-based Determ of Prolif Rate & Obser MR Imaging Featu (i.e., Ktrans or Microvas Permeabil; fBV, Tiss Fract Blood Vol), as Well With Spatially Reg Histolog Meas of Tum Cell Prolif (Ki67) & Microvas Density (CD31) at Corres Locat.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 18F-FLT PET Scan
Number analyzed (Participants) | 0

2. Secondary Outcome: Attempt to Corroborate Voxel-based Parameter Estimates Reflecting Tumor Cell Proliferation With Estimates Derived Using Standard ROI-based Pharmaco Modeling Methods, for Improving the Characterization of High-grade Gliomas Using Dynamic 18F-FLT PET-CT.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 18F-FLT PET Scan
Number analyzed (Participants) | 0

3. Secondary Outcome: Assess Whether Static Meas of 18F-FLT Uptake Can Ade Serve as Non-invasive Biomarker of Prolif Act or Whether Parametric Images, Based on Compart Analys of FLT Pharmas, Are Req by Correl Find of Both Appro With Region Histol Assays of Tum Cell Prolife.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 18F-FLT PET Scan
Number analyzed (Participants) | 0

4. Secondary Outcome: Evaluate Whether Differ in Gene Expression Seen Between Areas of Increas & Decreas Proliferative Activity on Parametric Maps Define Consistent Differential Transcriptome Signatures for Comparison With Known Molecular Subclasses of GBM & Known Pathways.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 18F-FLT PET Scan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 18F-FLT PET Scan
All-Cause Mortality (participants affected / at risk) | 11/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT00979810/Prot_SAP_000.pdf